CLINICAL TRIAL: NCT02752308
Title: Effectiveness of Caudal Epidural Block on Intraoperative Blood Loss During Hypospadias Repair; A Randomized Clinical Trial
Brief Title: Effectiveness of Caudal Epidural Block on Intraoperative Blood Loss During Hypospadias Repair
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Farshid Alizadeh, Associate Professor, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 393854
Record Dates: First submitted 2016-04-20; First posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias | interventions — Bupivacaine; Anesthesia, General; Fentanyl; Glucose; Sodium Chloride; Neostigmine; Atropine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- General anesthesia + caudal block (Active Comparator): Patients who receive general anesthesia plus caudal epidural block and dilute epinephrine injection before hypospadias repair, intraoperative fentanyl, intraoperative intravenous fluid and reversing the muscle relaxants' effect at the end of operation
  Interventions: Drug: Bupivacaine; Drug: Dilute epinephrine injection; Drug: Fentanyl; Drug: dextrose plus sodium chloride.; Drug: neostigmine and atropine; Procedure: Hypospadias repair
- General anesthesia only (Active Comparator): Patients who receive only general anesthesia and dilute epinephrine injection before hypospadias repair, intraoperative fentanyl, intraoperative intravenous fluid and reversing the muscle relaxants' effect at the end of operation
  Interventions: Procedure: General anesthesia; Drug: Dilute epinephrine injection; Drug: Fentanyl; Drug: dextrose plus sodium chloride.; Drug: neostigmine and atropine; Procedure: Hypospadias repair

INTERVENTIONS:
Drug: Bupivacaine — Injection of Bupivacaine in the epidural space (0.25%, 0.33mg/Kg)
  Other Names: Caudal block
  Arms: General anesthesia + caudal block
Procedure: General anesthesia — Induction with thiopental sodium 5 mg/Kg, atracurium 0.4 mg/Kg and fentanyl 2 mcg/Kg and maintenance with isoflurane and a combination of oxygen and nitrous oxide
  Arms: General anesthesia only
Drug: Dilute epinephrine injection — Injection of 1/100000 epinephrine solution along all incision lines
Drug: Fentanyl — fentanyl 2 mcg /Kg that is repeated during surgery whenever the heart rate or blood pressure increased more than 20% of its baseline
Drug: dextrose plus sodium chloride. — Four mL/Kg/hr of 5% dextrose plus 0.04 mL/Kg/hr of 20% sodium chloride. Each mL of blood loss was replaced by 3 ml of Ringer's solution
Drug: neostigmine and atropine — Injection of 0.04 mg/Kg of neostigmine and 0.02 mg/Kg of atropine, intravenously at the end of operation.
Procedure: Hypospadias repair — Surgical repair of hypospadias, using tubularized incised plate technique

SUMMARY:
From September 2014 to March 2015, 57 consecutive patients with hypospadias who are candidate for surgery will be enrolled in this randomized clinical trial.

Regional ethics committee of Isfahan University of Medical Sciences approved the protocol of the study and all parents will sign a written informed consent.

Inclusion criteria are age between 6 months to 15 years and hypospadias with any severity. Exclusion criteria are coagulopathy, history of previous failed surgery, skin infection , parents' disagreement with the protocol and any cardiac problem that made epinephrine injection contraindicated.

All selected patients will randomly allocate to one of the two groups: group A will receive caudal epidural block (CEB) plus general anesthesia before surgery and group B will receive general anesthesia before surgery and CEB afterwards. The surgical procedures will be performed by a single pediatric urologist (FA). The surgical technique will be tubularized incised plate in all cases.

Intraoperative blood loss will be determined by weighing all surgical gauzes used during procedure with a digital scale measure to the nearest 0.01 gram, every 10 minutes to minimize the effect of water vaporization on gauzes weights.

In addition to blood loss, operation time, dose of fentanyl used during procedure and length of the urethral plate defect will be recorded for each patient by trained nurses.

Demographics and disease characteristics as well as operation details will be compared in the two studied groups.

ELIGIBILITY:
Inclusion Criteria:

age between 6 months to 15 years and hypospadias with any severity

Exclusion Criteria:

coagulopathy, history of previous failed surgery, skin infection , parents' disagreement with the protocol and any cardiac problem that made epinephrine injection contraindicated

Ages: 6 Months to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | During procedure
  The amount of blood loss during the operation

SECONDARY OUTCOMES:
Dose of fentanyl used | during the operation
operation time | during procedure

IPD SHARING:
Plan to Share IPD: No